CLINICAL TRIAL: NCT00842569
Title: ERP Study of Brain Electrophysiological Patterns in Obesity
Brief Title: Brain Electrophysiological Patterns in Obesity
Status: Completed | Type: Observational
Sponsor: Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other)
Responsible Party: Dr Emmanuel DISSE, Centre de Recherche en Nutrition Humaine Rhone-Alpe
Other Study IDs: CRNHRA-09-001
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Obesity
Keywords: obesity; cognitive process; reward; P300; ERP; Event-related potential during oddball paradigm; brain electrophysiological patterns; externalizing factor
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal weighted: BMI<25
- Obese: BMI>30

SUMMARY:
There is growing evidence of behavioural and neurobiological overlaps between obesity and drug abuse. Reduction of the amplitude of P300, a component of event-related potentials (ERP) elicited by an oddball paradigm, is an electrophysiological characteristic and a marker of vulnerability in substance abuse. We want to determine whether obesity is associated with such electrophysiological features during an auditory oddball paradigm. We postulate that obesity could be associated with electrophysiological abnormalities that could be viewed as a possible vulnerability marker for food addiction.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the study are men and women aged 20-60 years, BMI 18.5-24.9 kg/m2 for control subjects and BMI>30 kg/m2 for obese subjects, stable body weight over the previous 3 months, report of sedentary or moderate physical activity

Exclusion Criteria:

* The exclusion criteria are pregnancy, post-menopausal women, any physiological or psychological illness that could influence the results, subjects likely to take medical drugs interfering with the electrophysiological parameters of the study, diabetes, hearing disorder, intense physical activity and report or evidence of excessive alcohol consumption, depressive state or eating disorders according to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: a healthy but normal-weighted or obese population. Depressive state or eating disorders were carefully evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of amplitudes and latencies of the P300 complex of Event Related Potential during an oddball paradigm, in normal-weighted and obese subjects

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel DISSE, MD, Principal Investigator — CRNH Rhone-Alpes
Locations (1):
- Centre de Recherche en Nutrition Humaine Rhone Alpes, Lyon, France

REFERENCES:
- [Background] Bauer LO, Hesselbrock VM. P300 decrements in teenagers with conduct problems: implications for substance abuse risk and brain development. Biol Psychiatry. 1999 Jul 15;46(2):263-72. doi: 10.1016/s0006-3223(98)00335-7. PMID 10418702
- [Background] Patrick CJ, Bernat EM, Malone SM, Iacono WG, Krueger RF, McGue M. P300 amplitude as an indicator of externalizing in adolescent males. Psychophysiology. 2006 Jan;43(1):84-92. doi: 10.1111/j.1469-8986.2006.00376.x. PMID 16629688
- [Background] Yoon HH, Iacono WG, Malone SM, McGue M. Using the brain P300 response to identify novel phenotypes reflecting genetic vulnerability for adolescent substance misuse. Addict Behav. 2006 Jun;31(6):1067-87. doi: 10.1016/j.addbeh.2006.03.036. Epub 2006 Apr 27. PMID 16644137